CLINICAL TRIAL: NCT00864851
Title: A Multi-Center, Open-Label, Randomized Study Evaluating the Safety and Efficacy of Three Dosing Regimens of Replagal Enzyme Replacement Therapy in Adult Patients With Fabry Disease
Brief Title: Safety and Efficacy Study of Several Replagal Dosing Regimens on Cardiac Function in Adults With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKT028; 2007-005543-22 (EudraCT Number)
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Replagal 0.2 mg/kg, IV, every other week (Active Comparator): Patients randomized to receive Replagal 0.2 mg/kg via intravenous infusion every other week for 52 weeks.
  Interventions: Biological: Replagal
- Replagal 0.2 mg/kg, IV, weekly (Active Comparator): Patients randomized to receive Replagal 0.2 mg/kg via intravenous infusion every week for 52 weeks.
  Interventions: Biological: Replagal
- Replagal 0.4 mg/kg, IV, weekly (Active Comparator): Patients randomized to receive Replagal 0.4 mg/kg via intravenous infusion every week for 52 weeks.
  Interventions: Biological: Replagal

INTERVENTIONS:
Biological: Replagal — Intravenous (IV) infusion for 12 months
  Other Names: algasidase alfa

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of various doses of Replagal in patients with cardiomyopathy due to Fabry disease.

DETAILED DESCRIPTION:
Fabry disease is an inherited, metabolic disease caused by mutations in the GALA gene. Patients with Fabry disease accumulate a complex glycosphingolipid named globotriaosylceramide (Gb3) in various tissues and organs. All organs are affected in Fabry disease but the majority of the morbidity and mortality are caused by cardiac, renal and neurological dysfunction. Accumulation of Gb3 in the heart causes hypertrophic cardiomyopathy, valvular abnormalities, arrhythmias and infarctions. Replagal has been shown to reduce Gb3 from key tissues and organs, and stabilize renal function in patients with Fabry disease. Evidence suggests that Replagal reduces left ventricular mass (LVM) and improves midwall fractional shortening (MFS) of the heart. Left ventricular hypertrophy is a major cause of morbidity and mortality in patients with Fabry disease.

This is a study of the safety and effectiveness of 3 dosing regimens of Replagal in adult patients with left ventricular hypertrophy due to Fabry disease.

The primary objective of the study is to compare the effects of 2 dosing regimens of Replagal (0.2 mg/kg IV every other week and 0.2 mg/kg IV weekly) on the reduction of left ventricular mass as measured by echocardiography.

The secondary objectives of this study are to compare the effects of 2 dosing regimens of Replagal (0.2 mg/kg IV every other week and 0.2 mg/kg IV weekly) on each of the following: exercise tolerance; improvement in disease-specific quality of life in heart failure patients; improvement of heart failure symptoms; magnitude of reduction in Gb3; rate of decline in renal function and improvement in the severity of proteinuria/albuminuria; and safety.

An alternative treatment regimen of 0.4 mg/kg Replagal IV weekly will also be explored but without formal comparison to the 0.2 mg/kg regimens. The investigation of the safety and efficacy of the 0.4 mg/kg IV weekly regimen is a secondary objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years-old;
* Male:Fabry disease confirmed by deficiency of alfa galactosidase A activity OR Female:Fabry disease confirmed by a mutation of the alfa galactosidase A gene;
* ERT-naïve;
* LVM/h > 50g/m2.7 for males and >47 g/m2.7 for females;
* Negative pregnancy test at enrollment and contraception use required throughout study for female patients;
* Signed informed consent;

Exclusion Criteria:

* Class IV heart failure;
* Clinically significant hypertension;
* Hemodynamically significant valvular stenosis or regurgitation;
* Morbid obesity;
* Known autosomal dominant sarcoplasmic contractile protein gene mutation;
* Treatment with any investigational drug or device within the 30 days;
* Unable to comply with the protocol as determined by the Investigator;
* Positive for hepatitis B, hepatitis C or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-12-29 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (4):
  - AKDHC Tucson Access Center, Tucson, Arizona
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - New York Unversity School of Medicine, New York, New York
  - O & O Alpan, LLC, Springfield, Virginia
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- The Charles University Hospital, Prague, Czechia
- Turku University Central Hospital, Turku, Finland
- Gobemador Irala y Coronel Lopez - Barrio Sojania, Asunción, Paraguay
- Poland (2):
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut Kardiologii, Warsaw
- General Hospital Slovenj Gradec, Slovenj Gradec, Slovenia
- Salford Royal NHS Foundation Trust, Salford, United Kingdom

REFERENCES:
- [Result] Malek LA, Chojnowska L, Spiewak M, Klopotowski M, Misko J, Petryka J, Milosz B, Ruzyllo W. Cardiac magnetic resonance imaging in patients with Fabry's disease. Kardiol Pol. 2010 Aug;68(8):929-34. PMID 20730727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Started | 20 | 19 | 5
Completed | 17 | 18 | 5
Not Completed | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Patient uncooperative | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Replagal 0.2 mg/kg, IV, Every Other Week: Patients who received Replagal 0.2 mg/kg via intravenous infusion every other week for 52 weeks.
- Replagal 0.2 mg/kg, IV, Weekly: Patients who received Replagal 0.2 mg/kg via intravenous infusion every week for 52 weeks.
- Replagal 0.4 mg/kg, IV, Weekly: Patients who received Replagal 0.4 mg/kg via intravenous infusion every week for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly | Total
Number analyzed (Participants) | 20 | 19 | 5 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (7.23) | 51.8 (11.42) | 49.4 (9.75) | 50.8 (9.34)
Age, Customized [Count of Participants; unit: Participants]
  18 to <45 years | 5 | 6 | 1 | 12
  >=45 years | 15 | 13 | 4 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 3 | 18
  Male | 14 | 10 | 2 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 19 | 18 | 5 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 19 | 5 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Left Ventricular Mass Indexed to Height (LVMI) [Mean (Standard Deviation); unit: g/m^2.7] | 76.1 (22.8) | 82.6 (28.3) | 99.3 (46.2) | 81.5 (28.5)
Baseline Maximal Oxygen Consumption (VO2 max) at Peak Exercise [Mean (Standard Deviation); unit: mL/min/kg] — 0.2 mg/kg Every Other Week: n=19 0.2 mg/kg Weekly: n=16 0.4 mg/kg Weekly: n=4 Total: n=39
  mL/min/kg | 20.2 (6.20) | 22.6 (6.89) | 24.0 (11.69) | 21.6 (7.05)
Baseline Distance Walked in 6-Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: m] — 0.2 mg/kg Every Other Week: n=18 0.2 mg/kg Weekly: n=19 0.4 mg/kg Weekly: n=5 Total: n=42
  m | 459.6 (103.0) | 514.3 (87.3) | 530.7 (90.2) | 492.8 (97.0)
Baseline Minnesota Living with Heart Failure Questionnaire (MLHF-Q) Summary Score [Mean (Standard Deviation); unit: scores on a scale] — Quality of life (QoL) was evaluated using the MLHF-Q, version 2. The questionnaire is designed to assess the degree to which heart failure symptoms affect a patient's daily life. The summary score ranges from 0 to 105, with a score of 105 representing the highest adverse impact on a patient's QoL.
  scores on a scale | 37.0 (23.8) | 21.1 (21.0) | 19.6 (26.5) | 28.1 (23.8)
Baseline New York Heart Association (NYHA) Functional Class [Count of Participants; unit: Participants] — Class I: Cardiac disease without limitation of physical activity. Ordinary physical activity does not cause undue symptoms. Class II: Cardiac disease with slight limitation of physical activity. Comfortable at rest, but ordinary physical activity causes symptoms. Class III: Cardiac disease with marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes symptoms. Class IV: Cardiac disease and unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. Note: Symptoms include fatigue, palpitation or dyspnea
  Participants
    Class I | 6 | 10 | 2 | 18
    Class II | 11 | 9 | 2 | 22
    Class III | 3 | 0 | 1 | 4
    Class IV | 0 | 0 | 0 | 0
Baseline Plasma Globotriaosylceramide (GB3) [Mean (Standard Deviation); unit: nmol/ml] | 6.067 (3.388) | 5.652 (5.212) | 5.292 (1.865) | 5.800 (4.104)
Baseline Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 82.0 (34.1) | 78.1 (33.8) | 72.1 (31.2) | 79.2 (33.1)
Baseline Urinary Albumin/Creatinine (A/Cr) Ratio [Mean (Standard Deviation); unit: mg/g] | 313.4 (614.07) | 293.4 (521.23) | 298.2 (175.85) | 303.0 (532.27)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 12 in Left Ventricular Mass Indexed to Height (LVMI)
Description: Left ventricular mass (LVM) was measured through echocardiography.
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Mean (Standard Deviation); unit: g/m^2.7
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 15 | 18 | 5
g/m^2.7 | 3.2 (12.5) | 0.5 (15.8) | -10.3 (11.8)

2. Secondary Outcome: Change From Baseline to Month 12 in Maximal Oxygen Consumption (VO2 Max) at Peak Exercise
Description: Exercise tolerance as measured by VO2 max at peak exercise using the standard exponential exercise protocol (STEEP).
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 14 | 15 | 4
mL/min/kg | -2.0 (3.24) | -0.3 (4.76) | 2.2 (5.85)

3. Secondary Outcome: Change From Baseline to Month 12 in Distance Walked in 6-Minute Walk Test (6MWT)
Description: Exercise tolerance using the 6MWT was measured as the total distance walked in 6 minutes.
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 15 | 18 | 5
m | -10.4 (87.7) | 37.9 (70.5) | 24.7 (45.7)

4. Secondary Outcome: Change From Baseline to Month 12 in the Minnesota Living With Heart Failure Questionnaire (MLHF-Q) Summary Score
Description: Quality of life (QoL) was evaluated using the MLHF-Q, version 2. The questionnaire is designed to assess the degree to which heart failure symptoms affect a patient's daily life. The summary score ranges from 0 to 105, with a score of 105 representing the highest adverse impact on a patient's QoL.
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 17 | 17 | 5
scores on a scale | -3.1 (16.7) | 2.1 (11.5) | -8.6 (12.3)

5. Secondary Outcome: Change From Baseline to Month 12 in New York Heart Association (NYHA) Functional Class
Description: The NYHA functional classification system relates symptoms to everyday activities and the patient's quality of life. NYHA Classification - The Stages of Heart Failure: Class I (Mild): No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath). Class II (Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea. Class III (Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV (Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Number; unit: participants
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 17 | 18 | 5
participants
  Improved ≥ 1 NYHA Functional Class | 2 | 2 | 2
  Maintained NYHA Functional Class | 15 | 16 | 3

6. Secondary Outcome: Change From Baseline to Month 12 in Plasma Globotriaosylceramide (GB3)
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Mean (Standard Deviation); unit: nmol/ml
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 17 | 18 | 5
nmol/ml | -1.046 (2.256) | -2.132 (4.363) | -2.076 (1.248)

7. Secondary Outcome: Change From Baseline to Month 12 in Estimated Glomerular Filtration Rate (eGFR)
Description: Renal function was assessed by an evaluation of change from baseline to Month 12 in eGFR as calculated using the Modification of Diet for Renal Disease (MDRD) equation.
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 17 | 18 | 5
mL/min/1.73m^2 | -1.2 (12.2) | -3.3 (12.7) | -1.7 (9.9)

8. Secondary Outcome: Change From Baseline to Month 12 in Urinary Albumin/Creatinine (A/Cr) Ratio
Time Frame: Baseline, Month 12 (Week 53)
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly
Number analyzed (Participants) | 17 | 17 | 5
mg/g | 83.9 (624.82) | -54.1 (322.51) | -54.2 (294.86)

9. Secondary Outcome: Safety Evaluation
Description: Adverse events were collected throughout the study, from the time of informed consent to approximately 30 days post-final infusion.
Time Frame: 56 Weeks
Population: Intent to Treat (ITT) Population: All randomized patients who received at least 1 complete or partial dose of Replagal. Analyses were performed on the ITT population because it was identical to the safety population.
Measure: Number; unit: participants
Groups:
- Overall: Total of all reporting groups.
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly | Overall
Number analyzed (Participants) | 20 | 19 | 5 | 44
participants
  No adverse event (AE) | 1 | 2 | 0 | 3
  At least one AE | 19 | 17 | 5 | 41
  At least one study drug-related AE | 6 | 6 | 2 | 14
  At least one infusion-related AE | 5 | 4 | 2 | 11
  At least one severe or life-threatening AE | 8 | 4 | 0 | 12
  At least one serious AE (SAE) | 8 | 5 | 2 | 15
  At least one study drug-related SAE | 1 | 0 | 0 | 1
  Discontinued due to an AE | 0 | 0 | 0 | 0
  Deaths | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 56 Weeks
Description: Adverse events were collected throughout the study, from the time of informed consent to approximately 30 days post-final infusion.
Arm/Group | Replagal 0.2 mg/kg, IV, Every Other Week | Replagal 0.2 mg/kg, IV, Weekly | Replagal 0.4 mg/kg, IV, Weekly | Overall
Serious Adverse Events (participants affected / at risk) | 8/20 | 5/19 | 2/5 | 15/44
Other Adverse Events (participants affected / at risk) | 19/20 | 17/19 | 5/5 | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal 0.2 mg/kg, IV, Every Other Week (N=20) | Replagal 0.2 mg/kg, IV, Weekly (N=19) | Replagal 0.4 mg/kg, IV, Weekly (N=5) | Overall (N=44)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spastic paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Replagal 0.2 mg/kg, IV, Every Other Week (N=20) | Replagal 0.2 mg/kg, IV, Weekly (N=19) | Replagal 0.4 mg/kg, IV, Weekly (N=5) | Overall (N=44)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (11) | 0 (0) | 8 (13)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 6 (6)
Respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (13) | 7 (13) | 1 (13) | 13 (39)
Oedema peripheral (General disorders) | 1 (1) | 4 (5) | 1 (3) | 6 (9)
Pyrexia (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1) | 6 (7)
Chest pain (General disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (3) | 0 (0) | 3 (4)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Implant site paraesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Implant site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (8) | 0 (0) | 0 (0) | 1 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (6) | 0 (0) | 7 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 1 (1) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 0 (0) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (10) | 0 (0) | 3 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2) | 2 (4)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Bundle branch block right (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (4) | 1 (1) | 0 (0) | 2 (5)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dilatation atrial (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 4 (6) | 1 (2) | 7 (11)
Dizziness (Nervous system disorders) | 2 (6) | 3 (4) | 0 (0) | 5 (10)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 2 (3) | 5 (6)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperreflexia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hypoaethesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (5)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spastic paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 3 (9) | 0 (0) | 5 (13)
Dental caries (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 4 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (5) | 1 (1) | 8 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Cardiac murmur (Investigations) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Haematocrit decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Body temperature decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mean haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
QRS axis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary lipids present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Biliary dilataton (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial bridging (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other